CLINICAL TRIAL: NCT06783829
Title: A Phase I Study of Safety, Tolerability, Pharmacokinetics and Efficacy of SHR-4394 Injection in Subjects With Prostate Cancer
Brief Title: A Study of SHR-4394 Injection in Subjects With Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-4394-101
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR4394 (Experimental)
  Interventions: Drug: SHR4394

INTERVENTIONS:
Drug: SHR4394 — SHR4394

SUMMARY:
This is an open label, multi-center, multiple dose Phase I study to evaluate the safety, tolerability, pharmacokinetics and efficacy of SHR-4394 injection in subjects with prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18-85 years old, male;
2. ECOG score for physical condition is 0-1 points;
3. Expected survival period ≥ 6 months;
4. Prostate adenocarcinoma confirmed by histological or cytological examination;
5. Patients with at least one metastasis lesion;
6. Disease progression on or after the most-recent prior regimen;
7. Continuous treatment with luteinizing hormone releasing hormone analogues (LHRHa) or previous bilateral orchidectomy;
8. Testosterone was at castration level;
9. Adequate organ function.

Exclusion Criteria:

1. Received systemic anticancer treatments or clinical investigational drugs 4 weeks prior to the initiation of the study treatment;
2. Unresolved to CTCAE 5.0>=grade 2 toxicities from previous anticancer therapy;
3. Meningeal metastasis history or clinical symptoms of central nervous system metastasis;
4. Uncontrollable tumor-related pain;
5. Uncontrolled pleural effusion, pericardial effusion, or abdominal effusion with clinical symptoms;
6. Other serious concomitant disease;
7. Previous or co-existing malignancies;
8. History of severe hypersensitivity reactions to either the drug substances or inactive ingredients of SHR-4394;
9. Active hepatitis B or active hepatitis C;
10. Other inappropriate situation considered by the investigator.

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 3 weeks.
Maximal tolerable dose (MTD) | 3 weeks.
Adverse events (AEs) | Screening up to study completion, an average of 1 year.
Recommended phase II dose (RP2D) | Screening up to study completion, an average of 1 year.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to approximately 2 years.
Duration of response (DOR) | Up to approximately 2 years.
Disease control rate (DCR) | Up to approximately 2 years.
overall survival (OS) | Up to approximately 2 years.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided